CLINICAL TRIAL: NCT06523894
Title: EASE (brEAst Stereo Elderly): A Phase Ia/Ib Study of Stereotactic Ablative Irradiation as an Alternative to Surgery in Elderly and Comorbid Breast Cancer Subjects
Brief Title: Ablative SBRT in Elderly BC Patients
Acronym: EASE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Pelagia Tsoutsou, Head of Radiation Oncology Department, University Hospital, Geneva
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BASEC 2024-00824
Record Dates: First submitted 2024-07-12; First posted 2024-07-26 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: radiotherapy; SBRT; inoperable
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase Ia/Ib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 fraction SBRT (Experimental): Treated volume up to 40 cc. Dose escalation from 21 Gy to 23 Gy to 25 Gy every 3 patients if no dose-limiting toxicity (DLT).
  Interventions: Radiation: SBRT
- 3 fractions SBRT (Experimental): Treated volume up to 60 cc. Dose escalation from 11Gy/fraction to 13Gy/fraction to 14Gy/fraction every 3 patients if no dose-limiting toxicity (DLT).
  Interventions: Radiation: SBRT
- 5 fractions SBRT (Experimental): Treated volume up to 110 cc. Dose escalation from 8Gy/fraction to 9Gy/fraction to 10Gy/fraction every 3 patients if no dose-limiting toxicity (DLT).
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Adapted to tumor volume BC SBRT

SUMMARY:
Stereotactic body radiotherapy (SBRT) is a modern radiotherapy technique, through which extremely high doses of irradiation are delivered in a very precise manner, within a few fractions. SBRT is increasingly used into clinical practice because it can provide excellent local control, comparable to surgery, in many tumor locations, such as lung, liver or bone. Efforts to develop it for BC treatment are promising, as it is safe, convenient, and effective. To date, SBRT for BC has been developed as an alternative method of partial-breast irradiation (PBI) in the pre- or post-operative setting. Therefore, the doses tested are comparable to the conventional doses used with surgery although its potential as sole local treatment for BC remains unknown. Higher SBRT doses are expected to permit obtaining an ablative effect on tumor and be suitable as an alternative to surgery, but this hypothesis has yet to be tested.

The aim of the present study is to prove the feasibility of SBRT as an ablative treatment in early breast cancer (BC). The primary objective is to find the maximum tolerated dose of SBRT that can be safely administered in inoperable patients with BC, the majority of whom are elderly or oldest old.

The overall objective is to determine whether high precision, dose- and fractionation- adapted SBRT is feasible and safe in inoperable patients with BC. The dose and fractionation-adapted SBRT regimen permits to test feasibility in different tumor sizes.

The primary objective of this study is to establish the maximum tolerated dose (MTD) that can be delivered with a single or few (up to 5) fractions of SBRT in inoperable patients with BC.

DETAILED DESCRIPTION:
SBRT will be performed using appropriate LINACs (Truebeam®, Varian, Palo Alto, US or Cyberknife®, Accuray, Morges, Switzerland) with a volumetric arc technique (VMAT), or non-coplanal technique, depending on the treating device. The medical devices have a CE certification and will be used in the trial as stated in the CE-marked instructions for use.

The gross tumor volume (GTV), as visualized on computed tomography (CT) within clips/fiducials, when present, with a 1mm (Cyberknife®)- 3mm (TrueBeam®) isotropic margin will be treated with an adaptive fractionation, depending on its total volume within 1,3 or 5 fractions. An elective volume of 2 cm around the GTV (clinical target volume (CTV)), plus a 1mm (Cyberknife®)- 3mm (TrueBeam®) isotropic margin will be treated at constant doses by fractionation cohort. These planning target volumes (PTVs) will be cropped at 5mm to skin and chest wall. The principle of irradiating an "elective volume" around the GTV will be used in this study, as done by Vasmel et al. [3]. This is decided because uncertainties do exist concerning true micro- and macrometastatic extension around the tumor, as visualized in the CT and delineation of the tumor on injected CT scans is not expected to be sufficient for coverage of macro and micrometastatic disease. Breast MRI is concordant to tumor size, as evaluated in pathology, within 0.5 cm for 53% of patients [4]. Organs at risk will be defined according to international guidelines [5].

Enrolment will be performed within 1-8 weeks after discussion in the HUG Breast Cancer Multidisciplinary Tumor Board (MTB).

All patients diagnosed with BC in our Institution, presenting the aforementioned characteristics, are candidates for screening for participation in the study, and will be offered clip placement, when feasible, during diagnostic biopsy by the specialized radiologist. Screening criteria will be assessed by the radiologist and radiation oncologist at the time of diagnostic biopsy.

Pre-screened patients will be discussed at the Institutional BC MTB. Eligible patients will be considered for the study.

Treatment procedures Treatment planning: Treatment planning will be performed using appropriate TPS (Eclipse®, (Varian, Palo Alto, US) or Accuray Precision®), with relevant techniques of SBRT in order to provide dose-delivery optimizations respecting predefined criteria for target coverage and normal-tissue constraints.

Accuracy issues: Accuracy of target volume delineation and dose delivery are of outmost importance for both tumor control and toxicity avoidance, given the limited number of fractions delivered. Accuracy issues are further detailed in the protocol section 3.4.1.

Quality assurance: A quality assurance (QA) program accompanies this trial, consisting of review of treatment plans by the trial medical physicist and the coordinating investigator.

SBRT fractionation will be adapted to PTV-GTV and PTV-CTV final volumes. With increasing volumes, more fractions will be used, according to the algorithm presented below, representing the dose-adapted fractionation regimens. SBRT will be delivered with isoeffective doses: a single fraction of 21, 23, or 25 Gy on day 1 or in three fractions of 11, 13 or 14 Gy/fraction on days 1, 3 and 5 or in five fractions of 8 or 9 or 10 Gy/fraction on days 1, 3, 5, 7 and 9. Dose per adaptive regimen will be escalated every three patients if no DLT appears.

In addition, patients will undergo physical exams at each study visit and (Serious) Adverse Events ((S)AE)s will be recorded. Questionnaires will be given to patients at selected study visits to assess Quality of Life (QoL). Other study procedures include measure of vital signs, ECOG performance status and record of concomitant treatments and procedures at each study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 70 years
2. Histologically confirmed diagnosis of BC, any time before study enrollment.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 3.
4. Patient considered inoperable in multidisciplinary board decision or refusing surgery. Main criteria determining inoperability are inability to receive general anesthesia after anesthetics and/or surgical evaluation. Criteria described in the statement of American Society of Anesthesiologists (ASA) {, #4699} and American College of Surgeons Surgical risk calculators {, #4695} are usually addressed in the multidisciplinary discussion (Appendix ).
5. Presence of measurable disease in the breast, defined as a lesion that can be accurately measured in at least one dimension with imaging (ultrasound, CT or MRI). Disease in the axilla or internal mammary chain is allowed and will be treated at the discretion of the radiation oncologist. Regional disease is not considered in measurements of local response.
6. Primary tumor accessible to SBRT, as defined by treating radiation oncologist.
7. Neo-adjuvant systemic therapy is allowed.
8. Tumor size in planning computed tomography (CT) permitting SBRT delivery. SBRT appropriateness is defined by the treating radiation oncologist.
9. Multifocality (over two tumor foci within the same breast quadrant) is allowed, as long as the total treatment volumes remain suitable for SBRT, as defined by the treating radiation oncologist.
10. Total tumor treatment volume/ whole breast volume ratio not exceeding 30%.
11. Previous treatment for BC to the contralateral breast is allowed. Previous treatment to the same breast for other reason than BC is allowed.
12. Capacity of patient to collaborate for SBRT delivery.
13. Capacity of patient to understand and sign a written informed consent according to International Council for Harmonization (ICH)/Good Clinical Practice (GCP) regulations before registration.

Exclusion Criteria:

1. Prior surgery for the current diagnosis.
2. Prior whole or partial breast irradiation to the involved breast.
3. Absolute contraindication to RT, such as Li-Fraumeni syndrome.
4. Current participation and receipt of study therapy or previous participation in a study of an investigational agent and receipt of study therapy or used an investigation device within 4 weeks of the first day of treatment.
5. Not able to communicate meaningfully with investigator and site staff and/or incapable of discernment.
6. Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

   -

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 4 weeks
  Dose before the dose-level at which one or more dose-limiting toxicity (DLT) (any treatment-related toxicity equal or superior to Grade 3, according to CTCAE v5) occurs within 4 weeks after end of study treatment (EOT).

SECONDARY OUTCOMES:
Early and late toxicities | 2 years
  • Early (up to 3 months after treatment start) and late (over 3 months and up to 2 years after treatment start) rates of toxicities, as graded by CTCAE v5, other than a dose-limiting toxicity (DLT), possibly, probably or definitely related to delivered treatment.
Differential safety profile between arms | 2 years
  Toxicity rates, as graded by CTCAE v5, will be compared between the fractionation regimens.
Explorative: clinically relevant technical parameters of SBRT | 2 years
  Technical parameters of treatment planning/ dose delivery and dose-volume histogram (DVH) parameters will be associated to toxicity in order to identify potential associations and constraints' thresholds.
Efficacy o SBRT on local control | 2 years
  Non progression, described as: stable local disease (SD), shrinkage of treated tumor (partial response (PR)) in imaging, as classified by RECIST v1.1 criteria, will be considered as response to treatment. Imaging should be consistent within study for a given patient. Progressive disease (PD) by RECIST v1.1 will be considered as disease progression, therefore non-response.
Explorative: Time to local, regional and distant progression | 2 years
  Time from enrolment until any objective tumor progression locally (within breast), regionally (supraclavicular, axillary or internal mammary chain area) or distantly (anywhere in the body beyond regional).
Quality of life (QoL) before and after SBRT | 2 years
  QoL parameters in the treatment population before and after treatment delivery and at follow-up, using appropriate questionnaires (EORTC QLQ-C30, EORTC QLQ-B23).
Explorative: Association between QoL and SBRT arm | 2 years
  Delivered treatment, in particular the risk-adapted dose and fractionation regimen used with QoL parameters after treatment delivery and at follow-up, using appropriate questionnaires (EORTC QLQ-C30, EORTC QLQ-B23) will be evaluated for the adapted regimens.
  Esthetic outcomes will be evaluated a. clinically, by the radiation oncologist and b. by the patient. Photos will be taken before treatment start and at follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Pelagia Tsoutsou, Pr, Study Chair — Radiation Oncology Department, Geneva University Hospital
Locations (1):
- Radiation Oncology Department, Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No